CLINICAL TRIAL: NCT06057337
Title: Promoting Health and Reducing Risk Among Hispanic Sexual Minority Youth and Their Families
Brief Title: Families With Pride ("Familias Con Orgullo").
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Guillermo Prado, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20230372; 1R01MD017588-01A1 (NIH)
Record Dates: First submitted 2023-07-14; First posted 2023-09-28 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Depression; Drug Use
Keywords: randomized controlled trial; Hispanic sexual minority youth; parent-centered
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Families with Pride ("Familias con Orgullo") (Experimental): Participants in this group will receive the Families with Pride (Familias con Orgullo) intervention. The intervention consists of seven multi parent group sessions, three multi adolescent group sessions, and four family sessions (parents participant in a total of 11 sessions, adolescents participate in a total of seven sessions) that will be delivered by a facilitator to the parent-child dyad across 12 weeks.
  Interventions: Behavioral: Families with Pride ("Familias con Orgullo")
- Community Practice (No Intervention): In this condition, participants will not receive an intervention, only the standard of care services for up to 12 weeks.

INTERVENTIONS:
Behavioral: Families with Pride ("Familias con Orgullo") — Families with Pride (Familias con Orgullo) aims to prevent the co-occurring epidemics of drug use and depression in Hispanic sexual minority youth. It focuses on improving parent support for the adolescent, parent acceptance of the adolescent, family functioning (e.g., communication), and decreasing stress and sexual minority stress. The program consists of 11 weekly, in-person sessions: 7 parent group sessions, 3 concurrent adolescent group sessions, both lasting two hours, 4 family sessions lasting 1 hour in either Spanish or English, depending on participant language preference. In the parent group sessions, parents come together to foster social support, family functioning, and increase parental support and acceptance for the adolescent. In the adolescent sessions, adolescents build skills in confronting and managing stressors related to being a sexual minority.
  Arms: Families with Pride ("Familias con Orgullo")

SUMMARY:
This study will evaluate the effects of a parenting intervention for Hispanic sexual minority youth in preventing/reducing drug use and depressive symptoms. It will also examine whether the intervention improves parent social support for the adolescent, parent acceptance, family functioning, and whether it reduces general stress and stress associated with being a Hispanic sexual minority.

ELIGIBILITY:
Inclusion Criteria:

* Youth, 13 - 19, who report at least one of the following: a) identify as gay, lesbian, or bisexual, or b) reports same-sex sexual behavior.
* Adolescent has their disclosed their sexual minority status to at least one parent.
* Adolescent is of Hispanic immigrant origin, defined by having at least one parent that self-identifies as Hispanic (English and Spanish speaking Hispanics can participate in the study).
* Adolescent lives with an adult parent who is willing to participate.
* Family lives in South Florida

Exclusion Criteria:

* Adolescent identifies as transgender.
* Family plans to move out of South Florida during the study period

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Adolescent does not identify as transgender.
Enrollment: 306 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2029-12-28 (Estimated); Study Completion 2029-12-28 (Estimated)

PRIMARY OUTCOMES:
Change in depression symptoms | Baseline up to 30 months
  Change in depression symptoms will be assessed with the Center for Epidemiological Studies Depression Scale. Scores range from 0 to 60 with higher scores indicating the presence of more symptoms.
Change in frequency of drug use | Baseline up to 30 months
  Change in drug use will be reported as the number of days of use over the previous 90 days at each timepoint.
Change in quantity of drug use | Baseline up to 30 months
  Change in drug use will be reported as the amount of use over the previous 90 days at each timepoint.

SECONDARY OUTCOMES:
Change in unprotected sexual behavior | Baseline up to 30 months
  Change in unprotected sexual behavior will be reported as number of days of sex without a condom as reported over the last 90 days at each timepoint.
Change in Family Functioning as assessed by the Parenting Practices Questionnaire | Baseline up to 30 months
  Change in family functioning will be reported using nine items from the Parenting Practices Questionnaire . Response range varies based on questions, but most response items range from 0 to 4 with higher values indicating better parenting. Scores range from 0 to 36.
Change in Family Functioning as assessed by the Parent-Adolescent Communication Scale | Baseline up to 30 months
  Change in family functioning will be reported using the Parent-Adolescent Communication Scale. The Parent-Adolescent Communication Scale is a 20-item questionnaire with a total score ranging from 20 to 100 with higher scores indicating better communication.
Changes in Adolescent Stress as assessed by the Perceived Stress Scale | Baseline up to 30 months
  Change in adolescent stress will be reported using the Perceived Stress Scale. The Perceived Stress Scale is a 10-item measure with response items ranging from 0 to 4. Higher scores indicate more stress. Scores range from 0 to 40.
Changes in Parent Acceptance of Adolescents Sexual Orientation as assessed by the Perceived Parental Reactions Scale | Baseline up to 30 months
  Changes in parent acceptance of adolescents sexual orientation will be reported using the Perceived Parental Reactions Scale. The Perceived Parental Reactions Scale is a 32-item measure with responses ranging from 1 to 5. Higher scores indicate more negative perceptions of their parents' reactions, with scores ranging from 32 to 160.
Changes in Sexual Minority Stress as assessed by the Sexual Minority Adolescent Stress Scale | Baseline up to 30 months
  Change in adolescent sexual minority stress will be reported using the Sexual Minority Adolescent Stress Scale. The Sexual Minority Adolescent Stress Scale is a 54-item measure with higher scores indicating more sexual minority stress. Scores range from 1 to 54.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Prado, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lozano A, Estrada Y, Scott D, Tapia MI, Santos HP Jr, Carrico AW, Zolobczuk J, Manker A, Prado G. Familias con Orgullo: Study protocol for an efficacy study of a family-based intervention for Hispanic sexual minority youth. PLoS One. 2023 Dec 15;18(12):e0295683. doi: 10.1371/journal.pone.0295683. eCollection 2023. PMID 38100451